CLINICAL TRIAL: NCT01633554
Title: The Ability of Prediction of Fibrosis for ST-2 as a Non-invasive Marker in Chronic Hepatitis B
Brief Title: ST-2; a Non-invasive Fibrosis Marker for Chronic Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Hakkı KALKAN, MD, Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 24190708; IKalkan24190708 (Registry Identifier: IKalkan24190708)
Record Dates: First submitted 2012-07-01; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Sequela of Chronic Liver Disease
Keywords: ST-2, IL-33, prediction, fibrosis, hepatitis B
MeSH Terms: conditions — Fibrosis; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Chronic Hepatitis B Group: Patients with chronic hepatitis B
- Cirrhosis: Patients with liver cirrhosis
- Control Group: Control Group: Healthy Volunteers

SUMMARY:
IL-33 is a recently identified number of the IL-1 family. Hepatic over-expression of IL-33 has been recently linked to liver fibrosis. ST-2 exerts pro-inflammatory effects of IL-33. We aimed to determine ability of ST2 to predict fibrosis in chronic hepatitis B.

DETAILED DESCRIPTION:
ST-2 is an IL-1 receptor family member and exists in both a membrane-bound isoform and a soluble (sST2) isoform. It has a functional ligand (Interleukin-33) and via ST-2/IL-33 inflammation and immunity is regulated. Hepatic over-expression of IL-33 has been recently linked to liver fibrosis. ST-2 exerts pro-inflammatory effects of IL-33. We aimed to determine ability of ST2 to predict fibrosis in chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic hepatitis B or liver cirrhosis

Exclusion Criteria:

* Accompanying chronic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 Healthy Volunteers 45 patients with chronic hepatitis B 25 patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Türkiye Yüksek İhtisas Education and research Hospital, Altındağ, Ankara, Turkey (Türkiye)